CLINICAL TRIAL: NCT03895372
Title: A PHASE 2, RANDOMIZED, DOUBLE BLIND, PLACEBO-CONTROLLED, STUDY TO EVALUATE THE SAFETY AND EFFICACY OF PF-06826647 IN PARTICIPANTS WITH MODERATE TO SEVERE PLAQUE PSORIASIS
Brief Title: A Study to Evaluate Safety and Efficacy of PF-06826647 For Moderate To Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C2501004; 2018-004669-16 (EudraCT Number)
Record Dates: First submitted 2019-03-13; First posted 2019-03-29 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ropsacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PF-06826647 Drug Dose Level 1 (Experimental): Delivered orally for 16 weeks during the Investigational Treatment Period
  Interventions: Drug: PF-06826647 or Placebo
- PF-06826647 Placebo (Experimental): Delivered orally for 16 weeks during the Investigational Treatment Period
  Interventions: Drug: PF-06826647 or Placebo
- PF-06826647 Drug Dose Level 2 (Experimental): Delivered orally for 16 weeks during the Investigational Treatment Period
  Interventions: Drug: PF-06826647 or Placebo
- PF-06826647 Drug Dose Level 3 (Experimental): Delivered orally for 16 weeks during the Investigational Treatment Period then 24 weeks in Extension Period.
  Interventions: Drug: PF-06826647 or Placebo; Drug: PF-06826647
- PF-06826647 Drug Dose Level 4 (Experimental): Delivered orally for 16 weeks then for 24 weeks in Extension Period.
  Interventions: Drug: PF-06826647 or Placebo; Drug: PF-06826647

INTERVENTIONS:
Drug: PF-06826647 or Placebo — Delivered orally (tablet) once daily (QD) for 16 weeks during the Investigational Treatment Period
Drug: PF-06826647 — Delivered orally (tablet) once daily (QD) for 24 weeks during the Extension Period
  Arms: PF-06826647 Drug Dose Level 3; PF-06826647 Drug Dose Level 4

SUMMARY:
This multicenter study is being conducted to provide additional PF-06826647 safety and tolerability data, and to further explore the clinical efficacy of PF-06826647 in the treatment of moderate to severe plaque psoriasis. Additionally, the study is intended to enable selection of oral dose and dosing regimen for the future clinical development of PF-06826647.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 75 years.
* Participants with a diagnosis of plaque psoriasis (psoriasis vulgaris) for at least 6 months.
* Have a PASI score of 12 or greater AND a Physician Global Assessment score of 3 (moderate) or 4 (severe).
* Have plaque-type psoriasis covering at least 10 % of total body surface area (BSA).

Exclusion Criteria:

* Have non-plaque forms of psoriasis.
* Drug-induced psoriasis.
* Current active infection.
* Infected with Mycobacterium tuberculosis (TB).
* Have any history of malignancies.
* Require treatment with prohibited concomitant medications(s).
* Positive for hepatitis B or C, or human immunodeficiency virus (HIV).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (22):
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - Center for Dermatology and Plastic Surgery/CCT, Scottsdale, Arizona
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Kern Research. Inc., Bakersfield, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Imaging Healthcare Specialists, San Diego, California
  - Medderm Associates Dermatology, San Diego, California
  - University Clinical Trials, San Diego, California
  - Renstar Medical Research, Ocala, Florida
  - MidState Skin Institute, Ocala, Florida
  - Advanced Diagnostic Group, Orange Park, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Hamilton Research, LLC, Alpharetta, Georgia
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - DelRicht Research, Baton Rouge, Louisiana
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Arlington Research Center, Inc., Arlington, Texas
- Canada (8):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SKiN Health, Cobourg, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Centre Radiologique de l'Estrie, Sherbrooke, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Japan (6):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Seibo International Catholic Hospital, Shinjuku-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka
  - Tokyo Medical University Hospital, Tokyo
- Poland (7):
  - Malopolskie Centrum Medyczn, Krakow, Lesser Poland Voivodeship
  - MTZ Clinical Research Sp. z o.o., Warsaw, Masovian Voivodeship
  - Zdrowie Osteo-Medic s.c. L. i A. Racewicz, A. i J. Supronik, Bialystok, Podlaskie Voivodeship
  - SpecDerm Poznanska Sp. J., Bialystok
  - Prywatny Gabinet Dermatologiczny Elzbieta Klujszo, Kielce
  - Pratia MCM Krakow, Krakow
  - Tomasz Blicharski Lubelskie Centrum Diagnostyczne, Swidnik, Lubelskie

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2501004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included 2 treatment periods (16-week investigational treatment period and 24-week extension treatment period) followed by a 4-week follow-up. A total of 179 participants were enrolled and 178 participants were treated in investigational treatment period and 153 participants completed this period and entered the extension treatment period. A total of 130 participants completed the extension treatment period.
Pre-assignment Details: This was a Phase 2b, randomized, double blind, placebo controlled, parallel group, and multicenter study in participants with moderate to severe plaque psoriasis.
Groups:
- Placebo QD->PF-06826647 200 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received matching placebo (2*25 mg size placebo and 4*100 mg size placebo)once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 200 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 116 days in investigational treatment period and 187 days in extension treatment period.
- Placebo QD->PF-06826647 400 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received matching placebo (2*25 mg size placebo and 4*100 mg size placebo) once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 400 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 116 days in investigational treatment period and 176 days in extension treatment period.
- PF-06826647 50 mg QD->PF-06826647 200 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 50 mg once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 200 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 119 days in investigational treatment period and 182 days in extension treatment period.
- PF-06826647 50 mg QD->PF-06826647 400 mg QD Group: This study includes 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 50 mg once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 400 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 119 days in investigational treatment period and 183 days in extension treatment period.
- PF-06826647 100 mg QD->PF-06826647 200 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 100 mg once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 200 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 115 days in investigational treatment period and 171 days in extension treatment period.
- PF-06826647 100 mg QD->PF-06826647 400 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 100 mg once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 400 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 115 days in investigational treatment period and 174 days in extension treatment period.
- PF-06826647 200 mg QD->PF-06826647 200 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 200 mg once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 200 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 120 days in investigational treatment period and 186 days in extension treatment period.
- PF-06826647 400 mg QD->PF-06826647 400 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 400 mg once a day (QD) in the investigational treatment period (16 weeks) and PF-06826647 400 mg QD in the extension treatment period (24 weeks). The maximum duration of treatment was 119 days in investigational treatment period and 180 days in extension treatment period.
Period: Investigational Treatment Period
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Started | 23 | 22 | 11 | 11 | 12 | 11 | 45 | 43
Completed | 19 | 19 | 10 | 9 | 12 | 9 | 37 | 38
Not Completed | 4 | 3 | 1 | 2 | 0 | 2 | 8 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 1 | 0 | 1 | 3 | 0
Period: Extension Treatment Period
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Started | 19 | 19 | 10 | 9 | 12 | 9 | 37 | 38
Completed | 16 | 14 | 10 | 8 | 9 | 8 | 33 | 32
Not Completed | 3 | 5 | 0 | 1 | 3 | 1 | 4 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 3
Not completed — Other | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were summarized by randomized treatment group for all randomized and treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group | Total
Number analyzed (Participants) | 23 | 22 | 11 | 11 | 12 | 11 | 45 | 43 | 178
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 9 | 11 | 7 | 3 | 6 | 6 | 24 | 20 | 86
  45-64 Years | 12 | 9 | 4 | 6 | 6 | 4 | 19 | 20 | 80
  >=65 Years | 2 | 2 | 0 | 2 | 0 | 1 | 2 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 2 | 5 | 3 | 4 | 19 | 8 | 56
  Male | 16 | 14 | 9 | 6 | 9 | 7 | 26 | 35 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 4 | 9
  Not Hispanic or Latino | 22 | 21 | 10 | 11 | 11 | 11 | 44 | 39 | 169
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 19 | 10 | 11 | 10 | 11 | 37 | 40 | 158
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Asian | 3 | 2 | 1 | 0 | 2 | 0 | 6 | 2 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI 90) Response Up to Week 16 - Investigational Treatment Period
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percentage of body surface area (BSA) affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 90 response was defined as at least a 90% reduction in PASI relative to baseline. The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: The analysis population included all randomized participants who received at least 1 dose of investigational product (PF-06826647 or placebo) after non-responder imputation applied (the participants discontinued due to coronavirus disease 2019 were removed).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received matching placebo (2*25 mg size placebo and 4*100 mg size placebo) once a day (QD) in the investigational treatment period (16 weeks). The maximum duration of treatment was 116 days in investigational treatment period.
- PF-06826647 50 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 50 mg once a day (QD) in the investigational treatment period (16 weeks). The maximum duration of treatment was 119 days in investigational treatment period.
- PF-06826647 100 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 100 mg once a day (QD) in the investigational treatment period (16 weeks). The maximum duration of treatment was 115 days in investigational treatment period.
- PF-06826647 200 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 200 mg once a day (QD) in the investigational treatment period (16 weeks). The maximum duration of treatment was 120 days in investigational treatment period.
- PF-06826647 400 mg QD Group: This study included 2 treatment periods: 16-week investigational treatment period and 24-week extension treatment period. The enrolled participants entered the investigational treatment period first and then the participants who completed the investigational treatment period entered the extension treatment period. The participants in this group received PF-06826647 400 mg once a day (QD) in the investigational treatment period (16 weeks). The maximum duration of treatment was 119 days in investigational treatment period.
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percentage of participants
  Week 1 | 0 [0.00 to 6.41] | 0 [0.00 to 12.60] | 0 [0.00 to 12.33] | 0 [0.00 to 5.97] | 0 [0.00 to 6.57]
  Week 2 | 0 [0.00 to 6.41] | 0 [0.00 to 12.60] | 0 [0.00 to 12.33] | 2.2 [0.23 to 9.17] | 0 [0.00 to 6.57]
  Week 4 | 0 [0.00 to 6.41] | 0 [0.00 to 12.60] | 0 [0.00 to 12.33] | 11.1 [5.50 to 21.80] | 7.3 [2.72 to 17.32]
  Week 6 | 0 [0.00 to 6.41] | 4.5 [0.48 to 19.56] | 4.8 [0.50 to 20.57] | 20.0 [11.72 to 31.73] | 26.8 [17.12 to 39.77]
  Week 8 | 2.4 [0.25 to 9.85] | 4.5 [0.48 to 19.56] | 4.8 [0.50 to 20.57] | 24.4 [15.47 to 35.88] | 34.1 [23.04 to 46.94]
  Week 12 | 2.4 [0.25 to 9.85] | 13.6 [5.12 to 31.13] | 9.5 [2.56 to 24.50] | 37.8 [25.96 to 50.95] | 48.8 [35.14 to 62.56]
  Week 16 | 4.8 [1.27 to 13.53] | 13.6 [5.12 to 31.13] | 9.5 [2.56 to 24.50] | 37.8 [25.96 to 50.95] | 51.2 [37.44 to 64.86]
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; p = 0.2621, Chan and Zhang method — One-sided Hochberg p-value, significant level is 0.05; Risk Difference (RD) = 8.87, 90% CI 2-sided [-4.50 to 26.26]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; p = 0.2621, Chan and Zhang method — One-sided Hochberg p-value, significant level is 0.05; Risk Difference (RD) = 4.76, 90% CI 2-sided [-7.07 to 21.48]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; p = 0.0004, Chan and Zhang method — One-sided Hochberg p-value, significant level is 0.05; Risk Difference (RD) = 33.02, 90% CI 2-sided [18.01 to 47.11]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; p < 0.0001, Chan and Zhang method — One-sided Hochberg p-value, significant level is 0.05; Risk Difference (RD) = 46.46, 90% CI 2-sided [30.62 to 60.56]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All-Causality), Week 16 to Week 40 - Extension Treatment Period
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. In this outcome measure, an AE was considered treatment-emergent if the event started on or after the first dosing day and time/start time but before the last dose plus the lag time.
Time Frame: From Week 16 to Week 40
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo) and who were treated in the extension treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 38
Participants
  Participants with AEs | 11 | 8 | 7 | 6 | 7 | 7 | 24 | 26
  Participants with SAEs | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
  Participants with severe AEs | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 3
  Participants discontinued from study due to AEs | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 3
  Participants discontinued study drug due to AE and continue study | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Participants with dose reduced or temporary discontinuation due to AEs | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 1

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment Related), Week 16 to Week 40 - Extension Treatment Period
Description: Treatment-related adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. In this outcome measure, an AE was considered treatment-emergent if the event started on or after the first dosing day and time/start time but before the last dose plus the lag time. Relatedness to investigational product (PF-06826647 or placebo) was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: From Week 16 to Week 40
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo) and who entered the extension treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 38
Participants
  Participants with AEs | 4 | 3 | 2 | 3 | 0 | 1 | 10 | 5
  Participants with SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Participants with severe AEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Participants discontinued from study due to AEs | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2
  Participants discontinued study drug due to AE and continue study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with dose reduced or temporary discontinuation due to AEs | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0

4. Primary Outcome: Number of Participants With Laboratory Test Abnormality - Hematology (Normal Baseline), Week 16 to Week 40 - Extension Treatment Period
Description: Following hematology parameters were analyzed for laboratory examination: hemoglobin (HGB), hematocrit, erythrocytes (Ery.), reticulocytes, Ery. mean corpuscular volume, Ery. mean corpuscular HGB, Ery. mean corpuscular HGB concentration, platelets, reticulocytes/erythrocytes, leukocytes, lymphocytes/leukocytes, neutrophils/leukocytes, basophils, basophils/leukocytes, eosinophils, eosinophils/leukocytes, monocytes, monocytes/leukocytes, activated partial thromboplastin time, prothrombin time, prothrombin international (Intl.) normalized ratio, neutrophils total count, and lymphocytes total count. LLN=lower limit of normal; ULN=upper limit of normal.
Time Frame: From Week 16 to Week 40
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo) and who were treated in the extension treatment period, with a normal baseline with at least one observation of the given laboratory test while on study treatment or during lag time from week 16 to week 40.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 38
Participants
  HGB (g/dL) <0.8*LLN: number analyzed (Participants) | 19 | 17 | 10 | 9 | 12 | 9 | 37 | 38
  HGB (g/dL) <0.8*LLN | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hematocrit (%) <0.8*LLN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 37
  Hematocrit (%) <0.8*LLN | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Erythrocytes (10^6/mm^3) <0.8*LLN: number analyzed (Participants) | 18 | 15 | 7 | 9 | 12 | 8 | 35 | 37
  Erythrocytes (10^6/mm^3) <0.8*LLN | 2 | 2 | 0 | 2 | 1 | 0 | 1 | 0
  Reticulocytes (10^3/mm^3) <0.5*LLN: number analyzed (Participants) | 19 | 17 | 10 | 9 | 11 | 8 | 34 | 36
  Reticulocytes (10^3/mm^3) <0.5*LLN | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Reticulocytes (10^3/mm^3) >1.5*ULN: number analyzed (Participants) | 19 | 17 | 10 | 9 | 11 | 8 | 34 | 36
  Reticulocytes (10^3/mm^3) >1.5*ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Ery. Mean Corpuscular Volume (um^3) <0.9*LLN: number analyzed (Participants) | 17 | 15 | 8 | 9 | 11 | 7 | 35 | 36
  Ery. Mean Corpuscular Volume (um^3) <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular Volume (um^3) >1.1*ULN: number analyzed (Participants) | 17 | 15 | 8 | 9 | 11 | 7 | 35 | 36
  Ery. Mean Corpuscular Volume (um^3) >1.1*ULN | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Ery. Mean Corpuscular HGB (pg/cell) <0.9*LLN: number analyzed (Participants) | 18 | 17 | 10 | 9 | 11 | 9 | 36 | 37
  Ery. Mean Corpuscular HGB (pg/cell) <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB (pg/cell) >1.1*ULN: number analyzed (Participants) | 18 | 17 | 10 | 9 | 11 | 9 | 36 | 37
  Ery. Mean Corpuscular HGB (pg/cell) >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (10^3/mm^3) <0.5*LLN: number analyzed (Participants) | 17 | 18 | 10 | 9 | 10 | 9 | 35 | 37
  Platelets (10^3/mm^3) <0.5*LLN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (10^3/mm^3) >1.75*ULN: number analyzed (Participants) | 17 | 18 | 10 | 9 | 10 | 9 | 35 | 37
  Platelets (10^3/mm^3) >1.75*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytes/Erythrocytes (%) <0.5*LLN: number analyzed (Participants) | 19 | 17 | 10 | 9 | 11 | 8 | 33 | 35
  Reticulocytes/Erythrocytes (%) <0.5*LLN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytes/Erythrocytes (%) >1.5*ULN: number analyzed (Participants) | 19 | 17 | 10 | 9 | 11 | 8 | 33 | 35
  Reticulocytes/Erythrocytes (%) >1.5*ULN | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2
  Leukocytes(10^3/mm^3) <0.6*LLN: number analyzed (Participants) | 18 | 18 | 10 | 7 | 11 | 9 | 35 | 35
  Leukocytes(10^3/mm^3) <0.6*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes(10^3/mm^3) >1.5*ULN: number analyzed (Participants) | 18 | 18 | 10 | 7 | 11 | 9 | 35 | 35
  Leukocytes(10^3/mm^3) >1.5*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes/Leukocytes (%) <0.8*LLN: number analyzed (Participants) | 18 | 18 | 10 | 6 | 11 | 8 | 30 | 36
  Lymphocytes/Leukocytes (%) <0.8*LLN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 18 | 18 | 10 | 6 | 11 | 8 | 30 | 36
  Lymphocytes/Leukocytes (%) >1.2*ULN | 0 | 5 | 0 | 0 | 0 | 0 | 2 | 5
  Neutrophils/Leukocytes (%) <0.8*LLN: number analyzed (Participants) | 18 | 18 | 10 | 6 | 10 | 8 | 32 | 37
  Neutrophils/Leukocytes (%) <0.8*LLN | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 3
  Neutrophils/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 18 | 18 | 10 | 6 | 10 | 8 | 32 | 37
  Neutrophils/Leukocytes (%) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 36 | 36
  Basophils (10^3/mm^3) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 16 | 18 | 10 | 8 | 11 | 8 | 33 | 31
  Basophils/Leukocytes (%) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 19 | 17 | 10 | 9 | 12 | 9 | 37 | 37
  Eosinophils (10^3/mm^3) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Eosinophils/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 19 | 18 | 9 | 9 | 12 | 9 | 35 | 36
  Eosinophils/Leukocytes (%) >1.2*ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 19 | 18 | 10 | 8 | 12 | 9 | 37 | 38
  Monocytes (10^3/mm^3) >1.2*ULN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Monocytes/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 37
  Monocytes/Leukocytes (%) >1.2*ULN | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Activated Partial Thromboplastin Time (sec) >1.1 x ULN | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Prothrombin Time (sec) >1.1*ULN: number analyzed (Participants) | 18 | 18 | 9 | 9 | 12 | 8 | 37 | 38
  Prothrombin Time (sec) >1.1*ULN | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Prothrombin Intl. Normalized Ratio >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils total count (10^3/mm^3) <0.8*LLN: number analyzed (Participants) | 19 | 18 | 10 | 7 | 10 | 9 | 31 | 35
  Neutrophils total count (10^3/mm^3) <0.8*LLN | 1 | 3 | 1 | 2 | 2 | 1 | 7 | 4
  Neutrophils total count (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 19 | 18 | 10 | 7 | 10 | 9 | 31 | 35
  Neutrophils total count (10^3/mm^3) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Lymphocytes total count (10^3/mm^3) <0.8*LLN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 11 | 9 | 37 | 38
  Lymphocytes total count (10^3/mm^3) <0.8*LLN | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocytes total count (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 11 | 9 | 37 | 38
  Lymphocytes total count (10^3/mm^3) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

5. Primary Outcome: Number of Participants With Laboratory Test Abnormality - Chemistry (Normal Baseline), Week 16 to Week 40 - Extension Treatment Period
Description: Following clinical chemistry parameters were analyzed for laboratory examination: bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase, protein, albumin, blood urea nitrogen, urea, creatinine, urate, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, triglycerides, sodium, potassium, chloride, calcium, bicarbonate, glucose, creatine kinase, and cholesterol.
Time Frame: From Week 16 to Week 40
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 38
Participants
  Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 18 | 18 | 10 | 9 | 12 | 8 | 35 | 38
  Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Direct Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 8 | 35 | 38
  Indirect Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (U/L) > 3.0*ULN: number analyzed (Participants) | 19 | 17 | 8 | 9 | 12 | 9 | 34 | 31
  Aspartate Aminotransferase (U/L) > 3.0*ULN | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
  Alanine Aminotransferase (U/L) > 3.0*ULN: number analyzed (Participants) | 18 | 16 | 7 | 8 | 11 | 8 | 33 | 25
  Alanine Aminotransferase (U/L) > 3.0*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Gamma Glutamyl Transferase (U/L) > 3.0*ULN: number analyzed (Participants) | 17 | 15 | 9 | 9 | 10 | 9 | 33 | 31
  Gamma Glutamyl Transferase (U/L) > 3.0*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Alkaline Phosphatase (U/L) > 3.0*ULN: number analyzed (Participants) | 17 | 17 | 9 | 8 | 11 | 9 | 35 | 38
  Alkaline Phosphatase (U/L) > 3.0*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) <0.8*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) <0.8*LLN: number analyzed (Participants) | 18 | 16 | 7 | 9 | 10 | 8 | 34 | 33
  Albumin (g/dL) <0.8*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) >1.2*ULN: number analyzed (Participants) | 18 | 16 | 7 | 9 | 10 | 8 | 34 | 33
  Albumin (g/dL) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (mg/dL) >1.3*ULN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 37
  Blood Urea Nitrogen (mg/dL) >1.3*ULN | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea (mg/dL) >1.3*ULN: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Urea (mg/dL) >1.3*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) >1.3*ULN: number analyzed (Participants) | 19 | 18 | 9 | 9 | 12 | 9 | 37 | 37
  Creatinine (mg/dL) >1.3*ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Urate (mg/dL) >1.2*ULN: number analyzed (Participants) | 17 | 17 | 9 | 9 | 12 | 9 | 34 | 38
  Urate (mg/dL) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  HDL Cholesterol (mg/dL) <0.8*LLN: number analyzed (Participants) | 16 | 15 | 9 | 8 | 9 | 8 | 33 | 32
  HDL Cholesterol (mg/dL) <0.8*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LDL Cholesterol (mg/dL) >1.2*ULN: number analyzed (Participants) | 16 | 14 | 10 | 8 | 9 | 8 | 33 | 30
  LDL Cholesterol (mg/dL) >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Triglycerides (mg/dL) >1.3*ULN: number analyzed (Participants) | 16 | 15 | 8 | 8 | 9 | 8 | 33 | 32
  Triglycerides (mg/dL) >1.3*ULN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Sodium (Meq/L) <0.95*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium (Meq/L) >1.05*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (Meq/L) <0.9*LLN: number analyzed (Participants) | 19 | 18 | 9 | 9 | 12 | 9 | 37 | 37
  Potassium (Meq/L) <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (Meq/L) >1.1*ULN: number analyzed (Participants) | 19 | 18 | 9 | 9 | 12 | 9 | 37 | 37
  Potassium (Meq/L) >1.1*ULN | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Chloride (Meq/L) <0.9*LLN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 37
  Chloride (Meq/L) <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride (Meq/L) >1.1*ULN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 37
  Chloride (Meq/L) >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) <0.9*LLN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 36 | 38
  Calcium (mg/dL) <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) >1.1*ULN: number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 36 | 38
  Calcium (mg/dL) >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bicarbonate (Meq/L) <0.9*LLN: number analyzed (Participants) | 19 | 17 | 9 | 9 | 12 | 9 | 37 | 37
  Bicarbonate (Meq/L) <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bicarbonate (Meq/L) >1.1*ULN: number analyzed (Participants) | 19 | 17 | 9 | 9 | 12 | 9 | 37 | 37
  Bicarbonate (Meq/L) >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) <0.6*LLN: number analyzed (Participants) | 10 | 13 | 7 | 6 | 10 | 6 | 19 | 25
  Glucose (mg/dL) <0.6*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) >1.5*ULN: number analyzed (Participants) | 10 | 13 | 7 | 6 | 10 | 6 | 19 | 25
  Glucose (mg/dL) >1.5*ULN | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2
  Creatine Kinase (U/L) >2.0*ULN: number analyzed (Participants) | 17 | 18 | 9 | 9 | 12 | 8 | 36 | 35
  Creatine Kinase (U/L) >2.0*ULN | 2 | 6 | 2 | 5 | 2 | 3 | 5 | 12
  Cholesterol (mg/dL) >1.3*ULN: number analyzed (Participants) | 15 | 14 | 9 | 7 | 9 | 8 | 30 | 32
  Cholesterol (mg/dL) >1.3*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Laboratory Test Abnormality - Urinalysis (Normal Baseline), Week 16 to Week 40 - Extension Treatment Period
Description: Following urinalysis parameters were analyzed for laboratory examination: urine pH, urine glucose, urine ketones, urine protein, urine hemoglobin, urine urobilinogen, urine bilirubin, urine nitrite, urine leukocyte esterase, urine erythrocytes, urine leukocytes, urine hyaline, and urine bacteria.
Time Frame: From Week 16 to Week 40
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 38
Participants
  Urine pH (Scalar) <4.5: number analyzed (Participants) | 16 | 13 | 10 | 8 | 9 | 8 | 33 | 32
  Urine pH (Scalar) <4.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine pH (Scalar) >8: number analyzed (Participants) | 16 | 13 | 10 | 8 | 9 | 8 | 33 | 32
  Urine pH (Scalar) >8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Glucose >=1: number analyzed (Participants) | 15 | 12 | 9 | 8 | 8 | 8 | 32 | 32
  Urine Glucose >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Ketones (Scalar) >=1: number analyzed (Participants) | 16 | 12 | 10 | 8 | 9 | 7 | 32 | 31
  Urine Ketones (Scalar) >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Protein >=1: number analyzed (Participants) | 16 | 13 | 10 | 8 | 9 | 8 | 33 | 32
  Urine Protein >=1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Urine Hemoglobin (Scalar) >=1: number analyzed (Participants) | 16 | 12 | 10 | 8 | 9 | 8 | 33 | 31
  Urine Hemoglobin (Scalar) >=1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Urine Urobilinogen (EU/dL) >=1: number analyzed (Participants) | 16 | 13 | 10 | 8 | 8 | 8 | 33 | 32
  Urine Urobilinogen (EU/dL) >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Urine Bilirubin (Scalar) >=1: number analyzed (Participants) | 16 | 13 | 10 | 8 | 9 | 8 | 33 | 32
  Urine Bilirubin (Scalar) >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Nitrite (Scalar) >=1: number analyzed (Participants) | 16 | 12 | 10 | 8 | 9 | 8 | 33 | 31
  Urine Nitrite (Scalar) >=1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Leukocyte Esterase (Scalar) >=1: number analyzed (Participants) | 15 | 12 | 10 | 7 | 9 | 8 | 32 | 32
  Urine Leukocyte Esterase (Scalar) >=1 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 0
  Urine Erythrocytes (Scalar) >=20: number analyzed (Participants) | 4 | 5 | 2 | 2 | 3 | 1 | 3 | 9
  Urine Erythrocytes (Scalar) >=20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Leukocytes (/HPF) >=20: number analyzed (Participants) | 4 | 4 | 2 | 1 | 3 | 1 | 8 | 14
  Urine Leukocytes (/HPF) >=20 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Hyaline Casts (/LPF) >1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urine Hyaline Casts (/LPF) >1 |  |  |  |  | 0 |  |  |
  Urine Bacteria (/LPF) >20: number analyzed (Participants) | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Urine Bacteria (/LPF) >20 | 0 |  |  | 0 |  |  | 0 |

7. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-defined Criteria, Week 16 to Week 40 - Extension Treatment Period
Description: Criteria for ECG abnormalities: maximum increase PR interval increase from baseline (IFB): percent change (Pctchg) >=25 percent (%) for baseline value of >200 milliseconds (msec) and Pctchg>=50% for baseline value of <=200 msec for PR interval, a maximum IFB: Pctchg>=50%, maximum QTcF interval (Fridericia's Correction) of 450 msec to <=480 msec, 480 msec to <=500 msec and a maximum change of <30 change =<60 or >60 msec from baseline.
Time Frame: From Week 16 to Week 40
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo) and were treated in the extension treatment period and evaluated against criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Number analyzed (Participants) | 17 | 17 | 10 | 9 | 11 | 8 | 37 | 36
Participants
  PR interval, single beat (msec) Pctchg >=25/50%: number analyzed (Participants) | 17 | 17 | 10 | 9 | 10 | 7 | 37 | 36
  PR interval, single beat (msec) Pctchg >=25/50% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  QRS duration, singe beat (msec) Pctchg >=50% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  QT interval, single beat (msec) >500 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  450< QTcF - Fridericia's correction formula (msec) <=480 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  480< QTcF - Fridericia's correction formula (msec) <=500 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  30< QTcF - Fridericia's correction formula (msec) change <=60 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 1
  QTcF - Fridericia's correction formula (msec) change >60 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Vital Sign Data Meeting Pre-defined Criteria, Week 16 to Week 40 - Extension Treatment Period
Description: The vital signs were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Criteria for vital signs abnormalities: sitting diastolic blood pressure (BP) < 50 millimeter of mercury (mmHg), sitting diastolic BP change >= 20 mmHg increase, sitting diastolic BP change >= 20 mmHg decrease, sitting systolic BP < 90 mmHg, sitting systolic BP change >= 30 mmHg increase, and sitting systolic BP change >= 30 mmHg decrease.
Time Frame: From Week 16 to Week 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
Number analyzed (Participants) | 19 | 18 | 10 | 9 | 12 | 9 | 37 | 38
Participants
  Sitting diastolic BP (mmHg) <50 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting diastolic BP (mmHg) change >= 20 increase | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 4
  Sitting diastolic BP (mmHg) change >= 20 decrease | 1 | 1 | 0 | 2 | 0 | 0 | 3 | 4
  Sitting systolic BP (mmHg) <90 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Sitting systolic BP (mmHg) change >= 30 increase | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 5
  Sitting systolic BP (mmHg) change >= 30 decrease | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1

9. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI 75) Response Up to Week 16 - Investigational Treatment Period
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least a 75 percent (%) reduction in PASI relative to Baseline. The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percentage of participants
  Week 1 | 0 [0.00 to 6.41] | 0 [0.00 to 12.60] | 0 [0.00 to 12.33] | 2.2 [0.23 to 9.17] | 0 [0.00 to 6.57]
  Week 2 | 4.8 [1.27 to 13.53] | 0 [0.00 to 12.60] | 0 [0.00 to 12.33] | 8.9 [3.93 to 18.01] | 2.4 [0.26 to 10.10]
  Week 4 | 7.1 [2.56 to 17.39] | 4.5 [0.48 to 19.56] | 0 [0.00 to 12.33] | 24.4 [15.47 to 35.88] | 31.7 [19.88 to 44.52]
  Week 6 | 7.1 [2.56 to 17.39] | 13.6 [5.12 to 31.13] | 4.8 [0.50 to 20.57] | 33.3 [21.80 to 46.08] | 43.9 [31.18 to 57.87]
  Week 8 | 4.8 [1.27 to 15.53] | 13.6 [5.12 to 31.13] | 14.3 [5.37 to 32.81] | 40.0 [28.66 to 52.89] | 61.0 [46.94 to 73.77]
  Week 12 | 9.5 [4.22 to 19.38] | 13.6 [5.12 to 31.13] | 9.5 [2.56 to 24.50] | 51.1 [38.26 to 64.12] | 70.7 [57.87 to 82.16]
  Week 16 | 14.3 [6.41 to 25.56] | 18.2 [8.17 to 35.25] | 9.5 [2.56 to 24.50] | 46.7 [33.79 to 59.13] | 73.2 [60.23 to 82.88]
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 3.90, 90% CI 2-sided [-11.82 to 23.42]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = -4.76, 90% CI 2-sided [-18.61 to 13.29]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 32.38, 90% CI 2-sided [14.32 to 47.52]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 58.89, 90% CI 2-sided [41.01 to 72.41]

10. Secondary Outcome: Percentage of Participants With Physician Global Assessment (PGA) of Psoriasis Score of "Clear" or "Almost Clear" and >=2 Points Improvement Up to Week 16 - Investigational Treatment Period
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percentage of participants
  Week 1 | 2.4 [0.25 to 9.85] | 0 [0.00 to 12.60] | 4.8 [0.50 to 20.57] | 4.4 [1.19 to 12.58] | 4.9 [1.30 to 13.87]
  Week 2 | 2.4 [0.25 to 9.85] | 0 [0.00 to 12.60] | 4.8 [0.50 to 20.57] | 11.1 [5.50 to 21.80] | 7.3 [2.72 to 17.32]
  Week 4 | 9.5 [4.22 to 19.38] | 9.1 [2.44 to 23.60] | 4.8 [0.50 to 20.57] | 35.6 [23.73 to 48.68] | 36.6 [24.57 to 50.00]
  Week 6 | 14.3 [6.41 to 25.56] | 13.6 [5.12 to 31.13] | 14.3 [5.37 to 32.81] | 46.7 [33.79 to 59.13] | 53.7 [39.77 to 66.11]
  Week 8 | 14.3 [6.41 to 25.56] | 18.2 [8.17 to 35.25] | 14.3 [5.37 to 32.81] | 44.4 [31.73 to 56.75] | 63.4 [50.00 to 75.43]
  Week 12 | 14.3 [6.41 to 25.56] | 18.2 [8.17 to 35.25] | 19.0 [8.58 to 37.19] | 46.7 [33.79 to 59.13] | 78.0 [64.86 to 87.04]
  Week 16 | 16.7 [9.06 to 27.68] | 18.2 [8.17 to 35.25] | 14.3 [5.37 to 32.81] | 44.4 [31.73 to 56.75] | 70.7 [57.87 to 82.16]
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 1.52, 90% CI 2-sided [-14.52 to 20.77]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = -2.38, 90% CI 2-sided [-17.67 to 17.01]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 27.78, 90% CI 2-sided [8.86 to 43.26]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 54.07, 90% CI 2-sided [36.46 to 68.27]

11. Secondary Outcome: Percentage of Participants With Physician Global Assessment (PGA) of Psoriasis Score of "Clear" or "Almost Clear", Up to Week 16 - Investigational Treatment Period
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percentage of participants
  Week 1 | 2.4 [0.25 to 9.85] | 0 [0.00 to 12.60] | 4.8 [0.50 to 20.57] | 4.4 [1.19 to 12.58] | 4.9 [1.30 to 13.87]
  Week 2 | 2.4 [0.25 to 9.85] | 0 [0.00 to 12.60] | 4.8 [0.50 to 20.57] | 11.1 [5.50 to 21.80] | 7.3 [2.72 to 17.32]
  Week 4 | 9.5 [4.22 to 19.38] | 9.1 [2.44 to 23.60] | 4.8 [0.50 to 20.57] | 35.6 [23.73 to 48.68] | 36.6 [24.57 to 50.00]
  Week 6 | 14.3 [6.41 to 25.56] | 13.6 [5.12 to 31.13] | 14.3 [5.37 to 32.81] | 46.7 [33.79 to 59.13] | 53.7 [39.77 to 66.11]
  Week 8 | 14.3 [6.41 to 25.56] | 18.2 [8.17 to 35.25] | 14.3 [5.37 to 32.81] | 44.4 [31.73 to 56.75] | 63.4 [50.00 to 75.43]
  Week 12 | 14.3 [6.41 to 25.56] | 18.2 [8.17 to 35.25] | 19.0 [8.58 to 37.19] | 46.7 [33.79 to 59.13] | 78.0 [64.86 to 87.04]
  Week 16 | 16.7 [9.06 to 27.68] | 18.2 [8.17 to 35.25] | 14.3 [5.37 to 32.81] | 44.4 [31.73 to 56.75] | 70.7 [57.87 to 82.16]
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 1.52, 90% CI 2-sided [-14.52 to 20.77]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = -2.38, 90% CI 2-sided [-17.67 to 17.01]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 27.78, 90% CI 2-sided [8.86 to 43.26]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 54.07, 90% CI 2-sided [36.46 to 68.27]

12. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 50 (PASI 50) Response Up to Week 16 - Investigational Treatment Period
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 50 response was defined as at least 50% reduction in PASI relative to Baseline.
Time Frame: Baseline up to Week 16
Population: The analysis population included all randomized participants who received at least 1 dose of investigational product (PF-06826647 or placebo) after non-responder imputation applied (the participants discontinued due to coronavirus disease 2019 were removed) and who were evaluated against criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percentage of participants
  Week 1: number analyzed (Participants) | 42 | 22 | 21 | 44 | 40
  Week 1 | 2.4 | 0 | 4.8 | 11.4 | 5.0
  Week 2 | 7.1 | 13.6 | 4.8 | 28.9 | 22.0
  Week 4: number analyzed (Participants) | 40 | 21 | 21 | 44 | 40
  Week 4 | 22.5 | 19.0 | 14.3 | 50.0 | 65.0
  Week 6: number analyzed (Participants) | 38 | 21 | 20 | 44 | 39
  Week 6 | 28.9 | 33.3 | 30.0 | 59.1 | 69.2
  Week 8: number analyzed (Participants) | 37 | 20 | 20 | 41 | 40
  Week 8 | 32.4 | 35.0 | 25.0 | 70.7 | 75.0
  Week 12: number analyzed (Participants) | 36 | 20 | 21 | 41 | 40
  Week 12 | 38.9 | 45.0 | 38.1 | 73.2 | 92.5
  Week 16: number analyzed (Participants) | 36 | 20 | 20 | 38 | 39
  Week 16 | 41.7 | 45.0 | 45.0 | 68.4 | 94.9

13. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 100 (PASI 100) Response Up to Week 16 - Investigational Treatment Period
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 100 response was defined as at least a 100 percent (%) reduction in PASI relative to Baseline.
Time Frame: Baseline up to Week 16
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percentage of participants
  Week 1: number analyzed (Participants) | 42 | 22 | 21 | 44 | 40
  Week 1 | 0 | 0 | 0 | 0 | 0
  Week 2 | 0 | 0 | 0 | 2.2 | 0
  Week 4: number analyzed (Participants) | 40 | 21 | 21 | 44 | 40
  Week 4 | 0 | 0 | 0 | 4.5 | 0
  Week 6: number analyzed (Participants) | 38 | 21 | 20 | 44 | 39
  Week 6 | 0 | 4.8 | 0 | 9.1 | 7.7
  Week 8: number analyzed (Participants) | 37 | 20 | 20 | 41 | 40
  Week 8 | 0 | 5.0 | 0 | 17.1 | 15.0
  Week 12: number analyzed (Participants) | 36 | 20 | 21 | 41 | 40
  Week 12 | 0 | 5.0 | 4.8 | 12.2 | 22.5
  Week 16: number analyzed (Participants) | 36 | 20 | 20 | 38 | 39
  Week 16 | 0 | 15.0 | 5.0 | 15.8 | 20.5

14. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Scores, Up to Week 16 - Investigational Treatment Period
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0= 0% to 6= 90-100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease. The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: The analysis population included all randomized participants who received at least 1 dose of investigational product (PF-06826647 or placebo) after non-responder imputation applied (the participants discontinued due to coronavirus disease 2019 were removed) and who had observed data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Units on a scale
  Week 1: number analyzed (Participants) | 42 | 22 | 21 | 44 | 40
  Week 1 | -1.88 (0.697) | -2.82 (0.969) | -1.96 (0.984) | -4.32 (0.676) | -3.00 (0.708)
  Week 2 | -3.44 (0.959) | -3.83 (1.330) | -3.24 (1.356) | -0.804 (0.926) | -7.40 (0.970)
  Week 4: number analyzed (Participants) | 40 | 21 | 21 | 44 | 40
  Week 4 | -5.08 (1.108) | -5.16 (1.528) | -4.68 (1.553) | -12.25 (1.065) | -12.16 (1.114)
  Week 6: number analyzed (Participants) | 38 | 21 | 20 | 44 | 39
  Week 6 | -6.02 (1.268) | -6.96 (1.737) | -7.53 (1.769) | -14.45 (1.212) | -14.78 (1.268)
  Week 8: number analyzed (Participants) | 37 | 20 | 20 | 41 | 40
  Week 8 | -7.43 (1.333) | -7.55 (1.827) | -9.29 (1.847) | -15.74 (1.274) | -17.12 (1.324)
  Week 12: number analyzed (Participants) | 36 | 20 | 21 | 41 | 40
  Week 12 | -8.09 (1.364) | -8.58 (1.863) | -10.02 (1.861) | -16.79 (1.300) | -19.69 (1.340)
  Week 16: number analyzed (Participants) | 36 | 20 | 20 | 38 | 39
  Week 16 | -7.88 (1.417) | -9.34 (1.932) | -11.42 (1.928) | -17.68 (1.354) | -20.21 (1.387)
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -1.46, 90% CI 2-sided [-5.42 to 2.51]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -3.54, 90% CI 2-sided [-7.50 to 0.42]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -9.80, 90% CI 2-sided [-13.05 to -6.56]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -12.33, 90% CI 2-sided [-15.61 to -9.04]

15. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Scores, Up to Week 16 - Investigational Treatment Period
Description: as for outcome 14
Time Frame: Baseline up to Week 16
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percent change
  Week 1: number analyzed (Participants) | 42 | 22 | 21 | 44 | 40
  Week 1 | -5.63 (2.858) | -9.42 (3.975) | -8.93 (4.039) | -17.41 (2.774) | -12.55 (2.908)
  Week 2 | -16.18 (3.809) | -14.80 (5.283) | -14.37 (5.385) | -33.65 (3.677) | -30.58 (3.851)
  Week 4: number analyzed (Participants) | 40 | 21 | 21 | 44 | 40
  Week 4 | -22.66 (4.437) | -20.88 (6.107) | -22.70 (6.205) | -51.26 (4.259) | -53.81 (4.449)
  Week 6: number analyzed (Participants) | 38 | 21 | 20 | 44 | 39
  Week 6 | -27.07 (4.833) | -30.25 (6.619) | -33.79 (6.739) | -60.63 (4.620) | -64.03 (4.828)
  Week 8: number analyzed (Participants) | 37 | 20 | 20 | 41 | 40
  Week 8 | -31.16 (4.983) | -33.27 (6.831) | -39.81 (6.909) | -66.51 (4.763) | -72.81 (4.954)
  Week 12: number analyzed (Participants) | 36 | 20 | 21 | 41 | 40
  Week 12 | -32.66 (5.137) | -37.24 (7.010) | -42.25 (6.996) | -70.28 (4.886) | -84.17 (5.039)
  Week 16: number analyzed (Participants) | 36 | 20 | 20 | 38 | 39
  Week 16 | -33.29 (5.369) | -41.92 (7.304) | -46.31 (7.271) | -74.03 (5.122) | -86.33 (5.236)
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -8.63, 90% CI 2-sided [-23.61 to 6.35]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -13.02, 90% CI 2-sided [-27.98 to 1.94]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -40.74, 90% CI 2-sided [-53.02 to -28.46]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -53.04, 90% CI 2-sided [-65.44 to -40.63]

16. Secondary Outcome: Change From Baseline in Peak-Pruritus Numerical Rating Scale (PP-NRS) Scores, Up to Week 16 - Investigational Treatment Period
Description: The intensity of pruritus was assessed by a PP-NRS, an 11-category numeric rating scale from 0 to 10, which was participant reported. Participants were asked to assess their itch over the past 24 hours, anchored by the terms "no itch" (0) and "worst itch imaginable" (10) at the ends. The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 38 | 17 | 20 | 42 | 38
Units on a scale
  Study Day 2, Week 1: number analyzed (Participants) | 38 | 17 | 19 | 41 | 37
  Study Day 2, Week 1 | -0.60 (0.238) | 0.05 (0.355) | -0.64 (0.331) | -0.76 (0.229) | -0.41 (0.241)
  Study Day 3, Week 1: number analyzed (Participants) | 38 | 17 | 20 | 40 | 38
  Study Day 3, Week 1 | -0.71 (0.239) | -0.65 (0.354) | -0.90 (0.325) | -0.83 (0.230) | -0.88 (0.239)
  Study Day 4, Week 1: number analyzed (Participants) | 38 | 17 | 19 | 41 | 37
  Study Day 4, Week 1 | -0.76 (0.234) | -0.83 (0.348) | -0.89 (0.323) | -1.24 (0.224) | -1.04 (0.236)
  Study Day 5, Week 1: number analyzed (Participants) | 38 | 16 | 18 | 41 | 35
  Study Day 5, Week 1 | -0.63 (0.233) | -0.91 (0.348) | -1.12 (0.324) | -1.26 (0.223) | -1.08 (0.237)
  Study Day 6, Week 1: number analyzed (Participants) | 38 | 17 | 19 | 41 | 34
  Study Day 6, Week 1 | -0.82 (0.246) | -0.94 (0.362) | -0.81 (0.336) | -1.49 (0.235) | -1.34 (0.250)
  Study Day 7, Week 1: number analyzed (Participants) | 37 | 17 | 18 | 38 | 37
  Study Day 7, Week 1 | -0.72 (0.272) | -1.11 (0.399) | -0.86 (0.372) | -1.75 (0.261) | -1.11 (0.273)
  Study Day 8, Week 1: number analyzed (Participants) | 37 | 16 | 20 | 42 | 37
  Study Day 8, Week 1 | -0.83 (0.274) | -1.26 (0.403) | -0.92 (0.371) | -1.65 (0.261) | -1.21 (0.276)
  Study Day 9, Week 1: number analyzed (Participants) | 37 | 17 | 18 | 39 | 37
  Study Day 9, Week 1 | -0.79 (0.289) | -1.32 (0.425) | -1.08 (0.394) | -1.50 (0.278) | -1.43 (0.292)
  Study Day 10, Week 1: number analyzed (Participants) | 37 | 16 | 20 | 40 | 36
  Study Day 10, Week 1 | -0.85 (0.284) | -1.48 (0.420) | -1.01 (0.384) | -1.63 (0.272) | -1.46 (0.286)
  Study Day 11, Week 1: number analyzed (Participants) | 33 | 15 | 19 | 37 | 36
  Study Day 11, Week 1 | -0.70 (0.291) | -1.55 (0.429) | -1.11 (0.392) | -1.67 (0.278) | -1.27 (0.291)
  Study Day 12, Week 2: number analyzed (Participants) | 32 | 16 | 18 | 38 | 35
  Study Day 12, Week 2 | -0.63 (0.289) | -1.67 (0.424) | -0.92 (0.390) | -1.93 (0.275) | -1.39 (0.289)
  Study Day 13, Week 2: number analyzed (Participants) | 34 | 16 | 19 | 41 | 33
  Study Day 13, Week 2 | -0.78 (0.294) | -1.49 (0.433) | -1.15 (0.397) | -2.18 (0.280) | -1.61 (0.296)
  Study Day 14, Week 2: number analyzed (Participants) | 34 | 17 | 20 | 38 | 36
  Study Day 14, Week 2 | -0.82 (0.317) | -1.66 (0.464) | -1.21 (0.426) | -2.15 (0.302) | -1.81 (0.317)
  Study Day 15, Week 2: number analyzed (Participants) | 36 | 16 | 19 | 40 | 38
  Study Day 15, Week 2 | -0.75 (0.308) | -1.48 (0.454) | -1.18 (0.417) | -2.20 (0.294) | -1.83 (0.309)
  Study Day 16, Week 2: number analyzed (Participants) | 34 | 16 | 18 | 37 | 37
  Study Day 16, Week 2 | -0.73 (0.314) | -1.52 (0.462) | -1.13 (0.426) | -2.29 (0.301) | -1.80 (0.314)
  Week 4: number analyzed (Participants) | 36 | 17 | 20 | 41 | 37
  Week 4 | -0.54 (0.354) | -1.74 (0.517) | -1.64 (0.477) | -2.90 (0.337) | -2.57 (0.354)
  Week 8: number analyzed (Participants) | 34 | 17 | 20 | 37 | 38
  Week 8 | -1.24 (0.391) | -1.10 (0.561) | -1.93 (0.517) | -4.10 (0.374) | -4.12 (0.381)
  Week 12: number analyzed (Participants) | 34 | 17 | 20 | 38 | 37
  Week 12 | -0.84 (0.455) | -1.66 (0.651) | -2.18 (0.599) | -3.92 (0.433) | -4.27 (0.442)
  Week 16: number analyzed (Participants) | 33 | 17 | 18 | 35 | 36
  Week 16 | -0.93 (0.453) | -2.15 (0.645) | -2.14 (0.604) | -4.40 (0.435) | -4.59 (0.440)
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -1.22, 90% CI 2-sided [-2.52 to 0.09]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -1.21, 90% CI 2-sided [-2.46 to 0.05]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -3.47, 90% CI 2-sided [-4.51 to -2.43]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -3.66, 90% CI 2-sided [-4.71 to -2.61]

17. Secondary Outcome: Percentage of Participants Achieving Psoriasis Symptom Inventory (PSI) Response of "Not at All" or "Mild" on Every Item, Up to Week 16 - Investigational Treatment Period
Description: The Psoriasis Symptom Inventory (PSI) is a self administered 8-item questionnaire that measures the severity of psoriasis symptoms over the past 24 hours and the past 7 days. The measure includes concepts of itch, pain, burning, stinging, cracking, scaling, flaking, and redness. Participants were asked to respond to each item using a 5-point Likert response scale: 0: not all severe, 1: mild, 2: moderate, 3: severe and 4: very severe. The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 42 | 22 | 21 | 45 | 41
Percentage of participants
  Study Day 2, Week 1 | 7.1 [2.65 to 17.39] | 0 [0.00 to 12.60] | 4.8 [0.50 to 20.57] | 6.7 [2.47 to 16.17] | 12.2 [6.05 to 23.04]
  Study Day 3, Week 1 | 7.1 [2.65 to 17.39] | 0 [0.00 to 12.60] | 19.0 [8.58 to 37.19] | 6.7 [2.47 to 16.17] | 12.2 [6.05 to 23.04]
  Study Day 4, Week 1 | 9.5 [4.22 to 19.38] | 4.5 [0.48 to 19.56] | 14.3 [5.37 to 32.81] | 13.3 [5.97 to 23.73] | 14.6 [6.57 to 26.23]
  Study Day 5, Week 1 | 7.1 [2.65 to 17.39] | 9.1 [2.44 to 23.60] | 14.3 [5.37 to 32.81] | 15.6 [8.42 to 25.96] | 19.5 [10.10 to 31.18]
  Study Day 6, Week 1 | 4.8 [1.27 to 13.53] | 13.6 [5.12 to 31.13] | 19.0 [8.58 to 37.19] | 20.0 [11.72 to 31.73] | 19.5 [10.10 to 31.18]
  Study Day 7, Week 1 | 9.5 [4.22 to 19.38] | 9.1 [2.44 to 23.60] | 19.0 [8.58 to 37.19] | 17.8 [9.17 to 29.70] | 19.5 [10.10 to 31.18]
  Study Day 8, Week 1 | 11.9 [5.91 to 22.74] | 9.1 [2.44 to 23.60] | 14.3 [5.37 to 32.81] | 20.0 [11.72 to 31.73] | 19.5 [10.10 to 31.18]
  Study Day 9, Week 1 | 9.5 [4.22 to 19.38] | 9.1 [2.44 to 23.60] | 9.5 [2.56 to 24.50] | 20.0 [11.72 to 31.73] | 22.0 [12.96 to 35.14]
  Study Day 10, Week 1 | 11.9 [5.91 to 22.74] | 4.5 [0.48 to 19.56] | 19.0 [8.58 to 37.19] | 24.4 [15.47 to 35.88] | 19.5 [10.10 to 31.18]
  Study Day 11, Week 1 | 9.5 [4.22 to 19.38] | 4.5 [0.48 to 19.56] | 19.0 [8.58 to 37.19] | 20.0 [11.72 to 31.73] | 26.8 [17.12 to 39.77]
  Study Day 12, Week 2 | 4.8 [1.27 to 13.53] | 4.5 [0.48 to 19.56] | 19.0 [8.58 to 37.19] | 22.2 [12.58 to 33.79] | 29.3 [17.84 to 42.13]
  Study Day 13, Week 2 | 11.9 [5.91 to 22.74] | 18.2 [8.17 to 32.25] | 14.3 [5.37 to 32.81] | 40.0 [28.66 to 52.89] | 26.8 [17.12 to 39.77]
  Study Day 14, Week 2 | 11.9 [5.91 to 22.74] | 22.7 [11.49 to 39.52] | 14.3 [5.37 to 32.81] | 33.3 [21.80 to 46.08] | 34.1 [23.04 to 46.94]
  Study Day 15, Week 2 | 4.8 [1.27 to 13.53] | 9.1 [2.44 to 23.60] | 14.3 [5.37 to 32.81] | 33.3 [21.80 to 46.08] | 29.3 [17.84 to 42.13]
  Study Day 16, Week 2 | 14.3 [6.41 to 25.56] | 13.6 [5.12 to 31.13] | 9.5 [2.56 to 24.50] | 24.4 [15.47 to 35.88] | 39.0 [26.23 to 53.06]
  Week 4 | 14.3 [6.41 to 25.56] | 13.6 [5.12 to 31.13] | 28.6 [13.24 to 46.41] | 44.4 [31.73 to 56.75] | 43.9 [31.18 to 57.87]
  Week 8 | 11.9 [5.91 to 22.74] | 22.7 [11.49 to 39.52] | 23.8 [12.06 to 41.72] | 53.3 [40.87 to 66.21] | 63.4 [50.00 to 75.43]
  Week 12 | 7.1 [2.65 to 17.39] | 31.8 [18.11 to 50.00] | 28.6 [13.24 to 46.41] | 55.6 [43.25 to 68.27] | 63.4 [50.00 to 75.43]
  Week 16 | 14.3 [6.41 to 25.56] | 27.3 [12.60 to 44.36] | 38.1 [20.57 to 58.28] | 55.6 [43.25 to 68.27] | 63.4 [50.00 to 75.43]
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 12.99, 90% CI 2-sided [-4.52 to 32.87]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 23.81, 90% CI 2-sided [2.62 to 44.64]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 41.27, 90% CI 2-sided [23.47 to 56.18]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Risk Difference (RD) = 49.13, 90% CI 2-sided [30.62 to 63.69]

18. Secondary Outcome: Change From Baseline in Psoriasis Symptom Inventory (PSI) Up to Week 16 - Investigational Treatment Period
Description: The Psoriasis Symptom Inventory (PSI) is a self administered 8-item questionnaire that measures the severity of psoriasis symptoms over the past 24 hours and the past 7 days. The measure includes concepts of itch, pain, burning, stinging, cracking, scaling, flaking, and redness. Participants were asked to respond to each item using a 5-point Likert response scale: 0: not all severe, 1: mild, 2: moderate, 3: severe and 4: very severe. The outcome of PSI is the sum of the scores for the 8 items. The total score range of PSI is 0-32. A negative change from baseline means a better outcome and the bigger score decrease means a better outcome. The statistical analysis was for the data at Week 16.
Time Frame: Baseline up to Week 16
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 38 | 18 | 21 | 42 | 39
Unit on a scale
  Study Day 2, Week 1: number analyzed (Participants) | 38 | 18 | 19 | 42 | 37
  Study Day 2, Week 1 | -1.51 (0.636) | -0.89 (0.927) | -1.98 (0.880) | -2.54 (0.605) | -1.25 (0.639)
  Study Day 3, Week 1: number analyzed (Participants) | 38 | 18 | 21 | 41 | 38
  Study Day 3, Week 1 | -2.70 (0.653) | -1.95 (0.952) | -3.65 (0.879) | -3.45 (0.624) | -2.79 (0.650)
  Study Day 4, Week 1: number analyzed (Participants) | 38 | 17 | 19 | 41 | 37
  Study Day 4, Week 1 | -2.88 (0.666) | -3.05 (0.985) | -3.95 (0.915) | -4.61 (0.637) | -4.28 (0.665)
  Study Day 5, Week 1: number analyzed (Participants) | 38 | 16 | 18 | 41 | 35
  Study Day 5, Week 1 | -2.55 (0.692) | -3.18 (1.032) | -3.87 (0.959) | -5.40 (0.661) | -3.93 (0.696)
  Study Day 6, Week 1: number analyzed (Participants) | 38 | 17 | 19 | 41 | 35
  Study Day 6, Week 1 | -3.01 (0.716) | -3.98 (1.058) | -3.94 (0.981) | -5.43 (0.684) | -4.77 (0.717)
  Study Day 7, Week 1: number analyzed (Participants) | 37 | 17 | 18 | 38 | 38
  Study Day 7, Week 1 | -3.23 (0.770) | -4.34 (1.134) | -4.08 (1.059) | -6.42 (0.740) | -4.90 (0.763)
  Study Day 8, Week 1: number analyzed (Participants) | 37 | 16 | 20 | 42 | 38
  Study Day 8, Week 1 | -3.27 (0.768) | -4.38 (1.137) | -4.65 (1.042) | -6.23 (0.731) | -5.67 (0.762)
  Study Day 9, Week 1: number analyzed (Participants) | 37 | 17 | 18 | 39 | 38
  Study Day 9, Week 1 | -3.11 (0.788) | -3.95 (1.159) | -4.54 (1.078) | -5.71 (0.756) | -5.70 (0.782)
  Study Day 10, Week 1: number analyzed (Participants) | 37 | 17 | 20 | 40 | 37
  Study Day 10, Week 1 | -3.29 (0.781) | -4.24 (1.150) | -4.15 (1.055) | -6.22 (0.747) | -6.02 (0.776)
  Study Day 11, Week 1: number analyzed (Participants) | 33 | 15 | 19 | 37 | 37
  Study Day 11, Week 1 | -2.89 (0.825) | -4.72 (1.216) | -4.41 (1.111) | -7.06 (0.787) | -6.03 (0.812)
  Study Day 12, Week 2: number analyzed (Participants) | 32 | 16 | 19 | 38 | 36
  Study Day 12, Week 2 | -3.04 (0.763) | -4.54 (1.118) | -4.65 (1.027) | -7.10 (0.726) | -6.62 (0.753)
  Study Day 13, Week 2: number analyzed (Participants) | 34 | 16 | 19 | 41 | 34
  Study Day 13, Week 2 | -2.94 (0.781) | -5.61 (1.149) | -4.79 (1.055) | -7.94 (0.742) | -7.16 (0.776)
  Study Day 14, Week 2: number analyzed (Participants) | 34 | 17 | 21 | 38 | 37
  Study Day 14, Week 2 | -3.25 (0.793) | -5.84 (1.162) | -5.22 (1.065) | -8.12 (0.757) | -7.09 (0.784)
  Study Day 15, Week 2: number analyzed (Participants) | 36 | 16 | 20 | 40 | 39
  Study Day 15, Week 2 | -2.71 (0.830) | -4.98 (1.227) | -5.23 (1.123) | -7.84 (0.793) | -7.47 (0.821)
  Study Day 16, Week 2: number analyzed (Participants) | 34 | 16 | 18 | 37 | 38
  Study Day 16, Week 2 | -3.27 (0.847) | -5.03 (1.250) | -4.83 (1.150) | -8.12 (0.810) | -7.45 (0.836)
  Week 4: number analyzed (Participants) | 36 | 17 | 20 | 41 | 38
  Week 4 | -2.53 (0.990) | -4.83 (1.449) | -6.58 (1.338) | -9.14 (0.943) | -9.02 (0.978)
  Week 8: number analyzed (Participants) | 34 | 17 | 20 | 37 | 39
  Week 8 | -3.45 (1.069) | -4.09 (1.536) | -7.30 (1.407) | -11.63 (1.022) | -12.19 (1.026)
  Week 12: number analyzed (Participants) | 34 | 17 | 20 | 38 | 38
  Week 12 | -2.27 (1.208) | -5.65 (1.722) | -7.35 (1.572) | -11.50 (1.146) | -13.42 (1.145)
  Week 16: number analyzed (Participants) | 33 | 17 | 18 | 35 | 37
  Week 16 | -1.87 (1.260) | -6.07 (1.782) | -8.31 (1.661) | -12.38 (1.205) | -12.68 (1.191)
Statistical Analysis 1: Comparison: Placebo QD Group vs PF-06826647 50 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -4.21, 90% CI 2-sided [-7.82 to -0.59]
Statistical Analysis 2: Comparison: Placebo QD Group vs PF-06826647 100 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -6.44, 90% CI 2-sided [-9.89 to -2.99]
Statistical Analysis 3: Comparison: Placebo QD Group vs PF-06826647 200 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -10.51, 90% CI 2-sided [-13.40 to -7.62]
Statistical Analysis 4: Comparison: Placebo QD Group vs PF-06826647 400 mg QD Group; The analysis was based on the data at Week 16; Test type: Superiority; Least Squares Mean Difference = -10.81, 90% CI 2-sided [-13.68 to -7.94]

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All-Causality), Up to Week 16 - Investigational Treatment Period
Description: as for outcome 2
Time Frame: Baseline up to Week 16
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 45 | 22 | 23 | 45 | 43
Participants
  Participants with AEs | 23 | 13 | 16 | 28 | 29
  Participants with SAEs | 0 | 1 | 0 | 1 | 0
  Participants with severe AEs | 1 | 0 | 1 | 2 | 3
  Participants discontinued from study due to AEs | 1 | 0 | 0 | 5 | 3
  Participants discontinued study drug due to AE and continue study | 0 | 0 | 0 | 1 | 0
  Participants with dose reduced or temporary discontinuation due to AEs | 1 | 1 | 2 | 3 | 3

20. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment Related), Up to Week 16 - Investigational Treatment Period
Description: Treatment-related adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug ((PF-06826647 or placebo). Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. In this outcome measure, an AE was considered treatment-emergent if the event started on or after the first dosing day and time/start time but before the last dose plus the lag time. Relatedness to investigational product (PF-06826647 or placebo) was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to Week 16
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 45 | 22 | 23 | 45 | 43
Participants
  Participants with AEs | 4 | 0 | 4 | 11 | 8
  Participants with SAEs | 0 | 0 | 0 | 1 | 0
  Participants with severe AEs | 0 | 0 | 0 | 2 | 1
  Participants discontinued from study due to AEs | 0 | 0 | 0 | 4 | 3
  Participants discontinued study drug due to AE and continue study | 0 | 0 | 0 | 1 | 0
  Participants with dose reduced or temporary discontinuation due to AEs | 0 | 0 | 0 | 1 | 1

21. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-defined Criteria, Up to Week 16 - Investigational Treatment Period
Description: Criteria for ECG abnormalities: Criteria for ECG abnormalities: maximum PR interval >=300 milliseconds (msec) and maximum increase PR interval increase from baseline (IFB): percent change (Pctchg) >=25 percent (%) for baseline value of >200 msec and Pctchg>=50% for baseline value of <=200 msec for PR interval, maximum QRS interval >=140 msec and a maximum IFB: Pctchg>=50%, maximum QTcF interval (Fridericia's Correction) of 450 msec to <=480 msec, 480 msec to <=500 msec and a maximum change of <30change<=60 or >60 msec from baseline.
Time Frame: Baseline up to Week 16
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo) and who had at least 1 ECG assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 44 | 22 | 23 | 44 | 43
Participants
  PR interval, single beat (msec) >=300 | 1 | 0 | 0 | 0 | 0
  PR interval, single beat (msec) Pctchg >=25/50% | 0 | 0 | 2 | 1 | 0
  QRS duration, single beat (msec) >=140 | 1 | 0 | 0 | 0 | 0
  QRS duration, single beat (msec) Pctchg >=50% | 1 | 0 | 1 | 0 | 0
  450< QTcF- Fridericia's correction formula (msec) <=480 | 1 | 0 | 2 | 2 | 0
  480< QTcF- Fridericia's correction formula (msec) <=500 | 1 | 0 | 0 | 0 | 0
  30< QTcF- Fridericia's correction formula (msec) change <=60 | 0 | 1 | 1 | 1 | 2
  QTcF- Fridericia's correction formula (msec) change >60 | 1 | 0 | 1 | 0 | 0

22. Secondary Outcome: Number of Participants With Vital Sign Data Meeting Pre-defined Criteria, Up to Week 16 - Investigational Treatment Period
Description: The vital signs were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Criteria for vital signs abnormalities: pulse rate >120 beats per minute (BPM), sitting diastolic blood pressure (BP) change >=20 millimeter of mercury (mmHg) increase, sitting diastolic BP change >=20 mmHg decrease, sitting systolic BP <90 mmHg, sitting systolic BP change >=30 mmHg increase, and sitting systolic BP change >=30 mmHg decrease.
Time Frame: Baseline up to Week 16
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo) and were evaluated against the criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 45 | 22 | 23 | 45 | 43
Participants
  Pulse rate (BMP) >120 | 0 | 0 | 0 | 0 | 1
  Sitting diastolic BP (mmHg) change >=20 increase: number analyzed (Participants) | 45 | 21 | 23 | 45 | 43
  Sitting diastolic BP (mmHg) change >=20 increase | 4 | 3 | 1 | 4 | 4
  Sitting diastolic BP (mmHg) change >=20 decrease: number analyzed (Participants) | 45 | 21 | 23 | 45 | 43
  Sitting diastolic BP (mmHg) change >=20 decrease | 4 | 2 | 0 | 2 | 4
  Sitting systolic BP (mmHg) <90 increase: number analyzed (Participants) | 45 | 21 | 23 | 45 | 43
  Sitting systolic BP (mmHg) <90 increase | 0 | 0 | 0 | 0 | 1
  Sitting systolic BP (mmHg) change >=30 increase: number analyzed (Participants) | 45 | 21 | 23 | 45 | 43
  Sitting systolic BP (mmHg) change >=30 increase | 0 | 1 | 2 | 2 | 2
  Sitting systolic BP (mmHg) change >=30 decrease: number analyzed (Participants) | 45 | 21 | 23 | 45 | 43
  Sitting systolic BP (mmHg) change >=30 decrease | 4 | 0 | 1 | 1 | 2

23. Secondary Outcome: Number of Participants With Laboratory Test Abnormality - Hematology (Normal Baseline), Up to Week 16 - Investigational Treatment Period
Description: Following hematology parameters were analyzed for laboratory examination: hemoglobin (HGB), hematocrit, erythrocytes (Ery.), reticulocytes, Ery. mean corpuscular volume, Ery. mean corpuscular HGB, Ery. mean corpuscular HGB concentration, platelets, reticulocytes/erythrocytes, leukocytes, lymphocytes/leukocytes, neutrophils/leukocytes, basophils, basophils/leukocytes, eosinophils, eosinophils/leukocytes, monocytes, monocytes/leukocytes, activated partial thromboplastin time, prothrombin time, neutrophils total count, and lymphocytes total count. LLN=lower limit of normal; ULN=upper limit of normal.
Time Frame: Baseline up to Week 16
Population: The analysis population included all participants who received at least 1 dose of investigational product (PF-06826647 or placebo), with a normal baseline with at least one observation of the given laboratory test while on study treatment or during lag time up to week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 45 | 22 | 23 | 45 | 43
Participants
  HGB (g/dL) <0.8*LLN: number analyzed (Participants) | 44 | 22 | 23 | 45 | 43
  HGB (g/dL) <0.8*LLN | 0 | 0 | 0 | 2 | 3
  Hematocrit (%) <0.8*LLN: number analyzed (Participants) | 45 | 22 | 23 | 45 | 42
  Hematocrit (%) <0.8*LLN | 0 | 0 | 0 | 2 | 3
  Erythrocytes (10^6/mm^3) <0.8*LLN: number analyzed (Participants) | 41 | 19 | 22 | 42 | 42
  Erythrocytes (10^6/mm^3) <0.8*LLN | 0 | 0 | 0 | 1 | 4
  Reticulocytes (10^3/mm^3) <0.5*LLN: number analyzed (Participants) | 44 | 22 | 21 | 42 | 41
  Reticulocytes (10^3/mm^3) <0.5*LLN | 0 | 0 | 0 | 0 | 2
  Reticulocytes (10^3/mm^3) >1.5*ULN: number analyzed (Participants) | 44 | 22 | 21 | 42 | 41
  Reticulocytes (10^3/mm^3) >1.5*ULN | 0 | 0 | 0 | 0 | 2
  Ery. Mean Corpuscular Volume (um^3) <0.9*LLN: number analyzed (Participants) | 38 | 18 | 20 | 43 | 41
  Ery. Mean Corpuscular Volume (um^3) <0.9*LLN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular Volume (um^3) >1.1*ULN: number analyzed (Participants) | 38 | 18 | 20 | 43 | 41
  Ery. Mean Corpuscular Volume (um^3) >1.1*ULN | 0 | 0 | 0 | 0 | 1
  Ery. Mean Corpuscular HGB (pg/cell) <0.9*LLN: number analyzed (Participants) | 43 | 22 | 22 | 44 | 42
  Ery. Mean Corpuscular HGB (pg/cell) <0.9*LLN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular Hemoglobin (pg/cell) >1.1*ULN: number analyzed (Participants) | 43 | 22 | 22 | 44 | 42
  Ery. Mean Corpuscular Hemoglobin (pg/cell) >1.1*ULN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9*LLN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1*ULN | 0 | 0 | 0 | 0 | 0
  Platelets (10^3/mm^3) <0.5*LLN: number analyzed (Participants) | 42 | 22 | 21 | 42 | 41
  Platelets (10^3/mm^3) <0.5*LLN | 0 | 0 | 0 | 0 | 1
  Platelets (10^3/mm^3) >1.75*ULN: number analyzed (Participants) | 42 | 22 | 21 | 42 | 41
  Platelets (10^3/mm^3) >1.75*ULN | 0 | 0 | 0 | 0 | 0
  Reticulocytes/Erythrocytes (%) <0.5*LLN: number analyzed (Participants) | 44 | 22 | 21 | 41 | 40
  Reticulocytes/Erythrocytes (%) <0.5*LLN | 0 | 0 | 0 | 0 | 2
  Reticulocytes/Erythrocytes (%) >1.5*ULN: number analyzed (Participants) | 44 | 22 | 21 | 41 | 40
  Reticulocytes/Erythrocytes (%) >1.5*ULN | 0 | 0 | 0 | 1 | 2
  Leukocytes(10^3/mm^3) <0.6*LLN: number analyzed (Participants) | 44 | 20 | 22 | 41 | 39
  Leukocytes(10^3/mm^3) <0.6*LLN | 0 | 0 | 0 | 1 | 1
  Leukocytes(10^3/mm^3) >1.5*ULN: number analyzed (Participants) | 44 | 20 | 22 | 41 | 39
  Leukocytes(10^3/mm^3) >1.5*ULN | 0 | 0 | 0 | 0 | 0
  Lymphocytes/Leukocytes (%) <0.8*LLN: number analyzed (Participants) | 44 | 19 | 21 | 37 | 39
  Lymphocytes/Leukocytes (%) <0.8*LLN | 0 | 1 | 0 | 1 | 3
  Lymphocytes/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 44 | 19 | 21 | 37 | 39
  Lymphocytes/Leukocytes (%) >1.2*ULN | 0 | 0 | 0 | 3 | 4
  Neutrophils/Leukocytes (%) <0.8*LLN: number analyzed (Participants) | 44 | 19 | 20 | 39 | 40
  Neutrophils/Leukocytes (%) <0.8*LLN | 1 | 0 | 0 | 2 | 2
  Neutrophils/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 44 | 19 | 20 | 39 | 40
  Neutrophils/Leukocytes (%) >1.2*ULN | 0 | 0 | 0 | 0 | 0
  Basophils (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 41
  Basophils (10^3/mm^3) >1.2*ULN | 0 | 0 | 0 | 1 | 0
  Basophils/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 42 | 21 | 21 | 41 | 36
  Basophils/Leukocytes (%) >1.2*ULN | 2 | 1 | 1 | 1 | 1
  Eosinophils (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 44 | 22 | 23 | 45 | 42
  Eosinophils (10^3/mm^3) >1.2*ULN | 1 | 1 | 0 | 0 | 0
  Eosinophils/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 45 | 21 | 23 | 43 | 41
  Eosinophils/Leukocytes (%) >1.2*ULN | 2 | 1 | 0 | 0 | 0
  Monocytes (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 45 | 21 | 23 | 45 | 42
  Monocytes (10^3/mm^3) >1.2*ULN | 1 | 0 | 1 | 0 | 0
  Monocytes/Leukocytes (%) >1.2*ULN: number analyzed (Participants) | 45 | 22 | 23 | 45 | 42
  Monocytes/Leukocytes (%) >1.2*ULN | 2 | 0 | 0 | 1 | 0
  Activated Partial Thromboplastin Time (sec) >1.1*ULN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 42
  Activated Partial Thromboplastin Time (sec) >1.1*ULN | 1 | 0 | 0 | 0 | 1
  Prothrombin Time (sec) >1.1*ULN: number analyzed (Participants) | 43 | 21 | 22 | 45 | 43
  Prothrombin Time (sec) >1.1*ULN | 1 | 0 | 0 | 0 | 3
  Neutrophils total count (10^3/mm^3) <0.8*LLN: number analyzed (Participants) | 45 | 20 | 21 | 38 | 39
  Neutrophils total count (10^3/mm^3) <0.8*LLN | 1 | 0 | 2 | 3 | 4
  Neutrophils total count (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 45 | 20 | 21 | 38 | 39
  Neutrophils total count (10^3/mm^3) >1.2*ULN | 3 | 1 | 1 | 2 | 2
  Lymphocytes total count (10^3/mm^3) <0.8*LLN: number analyzed (Participants) | 45 | 22 | 22 | 45 | 43
  Lymphocytes total count (10^3/mm^3) <0.8*LLN | 0 | 0 | 0 | 1 | 1
  Lymphocytes total count (10^3/mm^3) >1.2*ULN: number analyzed (Participants) | 45 | 22 | 22 | 45 | 43
  Lymphocytes total count (10^3/mm^3) >1.2*ULN | 0 | 0 | 1 | 1 | 1

24. Secondary Outcome: Number of Participants With Laboratory Test Abnormality - Chemistry (Normal Baseline), Up to Week 16 - Investigational Treatment Period
Description: Following clinical chemistry parameters were analyzed for laboratory examination: bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase, protein, albumin, blood urea nitrogen, urea, creatinine, urate, high-density lipoprotein (HDL) cholesterol, triglycerides, sodium, potassium, chloride, calcium, bicarbonate, glucose, creatine kinase, and cholesterol. LLN=lower limit of normal; ULN=upper limit of normal.
Time Frame: Baseline up to Week 16.
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 45 | 22 | 23 | 45 | 43
Participants
  Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 44 | 22 | 22 | 43 | 42
  Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 45 | 22 | 22 | 43 | 43
  Indirect Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (U/L) > 3.0*ULN: number analyzed (Participants) | 43 | 20 | 23 | 40 | 36
  Aspartate Aminotransferase (U/L) > 3.0*ULN | 1 | 0 | 1 | 0 | 0
  Alanine Aminotransferase (U/L) > 3.0*ULN: number analyzed (Participants) | 40 | 18 | 21 | 38 | 30
  Alanine Aminotransferase (U/L) > 3.0*ULN | 1 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase (U/L) > 3.0*ULN: number analyzed (Participants) | 38 | 21 | 21 | 41 | 36
  Gamma Glutamyl Transferase (U/L) > 3.0*ULN | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) > 3.0*ULN: number analyzed (Participants) | 41 | 20 | 22 | 43 | 43
  Alkaline Phosphatase (U/L) > 3.0*ULN | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) <0.8*LLN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 43
  Protein (g/dL) <0.8*LLN | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) >1.2*ULN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 43
  Protein (g/dL) >1.2*ULN | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) <0.8*LLN: number analyzed (Participants) | 40 | 19 | 20 | 41 | 38
  Albumin (g/dL) <0.8*LLN | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) >1.2*ULN: number analyzed (Participants) | 40 | 19 | 20 | 41 | 38
  Albumin (g/dL) >1.2*ULN | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (mg/dL) >1.3*ULN: number analyzed (Participants) | 45 | 22 | 23 | 45 | 42
  Blood Urea Nitrogen (mg/dL) >1.3*ULN | 1 | 0 | 0 | 2 | 0
  Urea (mg/dL) >1.3*ULN: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Urea (mg/dL) >1.3*ULN |  |  | 0 |  |
  Creatinine (mg/dL) >1.3*ULN: number analyzed (Participants) | 45 | 21 | 23 | 45 | 42
  Creatinine (mg/dL) >1.3*ULN | 0 | 0 | 0 | 1 | 1
  Urate (mg/dL) >1.2*ULN: number analyzed (Participants) | 40 | 20 | 23 | 41 | 43
  Urate (mg/dL) >1.2*ULN | 0 | 0 | 0 | 0 | 0
  HDL Cholesterol (mg/dL) <0.8*LLN: number analyzed (Participants) | 40 | 21 | 23 | 43 | 43
  HDL Cholesterol (mg/dL) <0.8*LLN | 0 | 0 | 0 | 0 | 0
  Triglycerides (mg/dL) >1.3*ULN: number analyzed (Participants) | 39 | 20 | 23 | 43 | 43
  Triglycerides (mg/dL) >1.3*ULN | 1 | 0 | 0 | 0 | 3
  Sodium (Meq/L) <0.95*LLN | 0 | 0 | 0 | 0 | 0
  Sodium (Meq/L) >1.05*ULN | 0 | 0 | 0 | 0 | 0
  Potassium (Meq/L) <0.9*LLN: number analyzed (Participants) | 45 | 21 | 23 | 45 | 41
  Potassium (Meq/L) <0.9*LLN | 0 | 0 | 0 | 0 | 0
  Potassium (Meq/L) >1.1*ULN: number analyzed (Participants) | 45 | 21 | 23 | 45 | 41
  Potassium (Meq/L) >1.1*ULN | 1 | 0 | 1 | 0 | 0
  Chloride (Meq/L) <0.9*LLN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 42
  Chloride (Meq/L) <0.9*LLN | 0 | 0 | 0 | 0 | 0
  Chloride (Meq/L) >1.1*ULN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 42
  Chloride (Meq/L) >1.1*ULN | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) <0.9*LLN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 43
  Calcium (mg/dL) <0.9*LLN | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) >1.1*ULN: number analyzed (Participants) | 45 | 22 | 23 | 44 | 43
  Calcium (mg/dL) >1.1*ULN | 0 | 0 | 0 | 0 | 0
  Bicarbonate (Meq/L) <0.9*LLN: number analyzed (Participants) | 44 | 21 | 23 | 45 | 42
  Bicarbonate (Meq/L) <0.9*LLN | 0 | 0 | 1 | 0 | 0
  Bicarbonate (Meq/L) >1.1*ULN: number analyzed (Participants) | 44 | 21 | 23 | 45 | 42
  Bicarbonate (Meq/L) >1.1*ULN | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) <0.6*LLN: number analyzed (Participants) | 29 | 16 | 18 | 25 | 27
  Glucose (mg/dL) <0.6*LLN | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) >1.5*ULN: number analyzed (Participants) | 29 | 16 | 18 | 25 | 27
  Glucose (mg/dL) >1.5*ULN | 1 | 0 | 0 | 0 | 1
  Creatine Kinase (U/L) >2.0*ULN: number analyzed (Participants) | 42 | 20 | 22 | 42 | 40
  Creatine Kinase (U/L) >2.0*ULN | 3 | 3 | 2 | 9 | 15
  Cholesterol (mg/dL) >1.3*ULN: number analyzed (Participants) | 38 | 20 | 23 | 38 | 43
  Cholesterol (mg/dL) >1.3*ULN | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Laboratory Test Abnormality - Urinalysis (Normal Baseline), Up to Week 16 - Investigational Treatment Period
Description: as for outcome 6
Time Frame: Baseline up to Week 16
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD Group | PF-06826647 50 mg QD Group | PF-06826647 100 mg QD Group | PF-06826647 200 mg QD Group | PF-06826647 400 mg QD Group
Number analyzed (Participants) | 45 | 22 | 23 | 45 | 43
Participants
  Urine pH (Scalar) <4.5: number analyzed (Participants) | 39 | 22 | 23 | 43 | 41
  Urine pH (Scalar) <4.5 | 0 | 0 | 0 | 0 | 0
  Urine pH (Scalar) >8: number analyzed (Participants) | 39 | 22 | 23 | 43 | 41
  Urine pH (Scalar) >8 | 0 | 0 | 0 | 0 | 0
  Urine Glucose >=1: number analyzed (Participants) | 37 | 21 | 22 | 42 | 41
  Urine Glucose >=1 | 0 | 0 | 0 | 1 | 1
  Urine Ketones (Scalar) >=1: number analyzed (Participants) | 38 | 22 | 22 | 40 | 40
  Urine Ketones (Scalar) >=1 | 2 | 0 | 1 | 0 | 2
  Urine Protein >=1: number analyzed (Participants) | 39 | 22 | 23 | 42 | 41
  Urine Protein >=1 | 1 | 0 | 0 | 1 | 2
  Urine Hemoglobin (Scalar) >=1: number analyzed (Participants) | 38 | 22 | 23 | 43 | 40
  Urine Hemoglobin (Scalar) >=1 | 3 | 1 | 0 | 4 | 0
  Urine Urobilinogen (EU/dL) >=1: number analyzed (Participants) | 39 | 22 | 22 | 43 | 40
  Urine Urobilinogen (EU/dL) >=1 | 1 | 0 | 0 | 1 | 2
  Urine Bilirubin (Scalar) >=1: number analyzed (Participants) | 39 | 22 | 23 | 43 | 41
  Urine Bilirubin (Scalar) >=1 | 0 | 0 | 0 | 0 | 0
  Urine Nitrite (Scalar) >=1: number analyzed (Participants) | 38 | 22 | 23 | 43 | 40
  Urine Nitrite (Scalar) >=1 | 0 | 1 | 0 | 0 | 0
  Urine Leukocyte Esterase (Scalar) >=1: number analyzed (Participants) | 37 | 21 | 23 | 41 | 41
  Urine Leukocyte Esterase (Scalar) >=1 | 1 | 2 | 0 | 1 | 0
  Urine Erythrocytes (Scalar) >=20: number analyzed (Participants) | 13 | 5 | 8 | 12 | 19
  Urine Erythrocytes (Scalar) >=20 | 1 | 0 | 0 | 1 | 0
  Urine Leukocytes (/HPF) >=20: number analyzed (Participants) | 12 | 6 | 8 | 18 | 18
  Urine Leukocytes (/HPF) >=20 | 1 | 0 | 0 | 0 | 0
  Urine Hyaline Casts (/LPF) >1: number analyzed (Participants) | 1 | 1 | 0 | 3 | 1
  Urine Hyaline Casts (/LPF) >1 | 1 | 1 |  | 3 | 1
  Urine Bacteria (/LPF) >20: number analyzed (Participants) | 2 | 1 | 1 | 4 | 0
  Urine Bacteria (/LPF) >20 | 0 | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment on Day 1 to 28 calendar days after the last dose of study treatment on Day 280
Description: Each AE was to be assessed to determine if it met the criteria for SAEs. If an SAE occurred, expedited reporting followed local and international regulations, as appropriate. In Section Outcome Measures, there were 2 separate summary data for the 2 periods is because the investigational treatment period contains the data for the primary endpoint.
Arm/Group | Placebo QD->PF-06826647 200 mg QD Group | Placebo QD->PF-06826647 400 mg QD Group | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/11 | 0/11 | 0/12 | 0/11 | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/22 | 0/11 | 1/11 | 0/12 | 1/11 | 3/45 | 0/43
Other Adverse Events (participants affected / at risk) | 14/23 | 11/22 | 10/11 | 8/11 | 9/12 | 9/11 | 29/45 | 32/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD->PF-06826647 200 mg QD Group (N=23) | Placebo QD->PF-06826647 400 mg QD Group (N=22) | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group (N=11) | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group (N=11) | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group (N=12) | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group (N=11) | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group (N=45) | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group (N=43)
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD->PF-06826647 200 mg QD Group (N=23) | Placebo QD->PF-06826647 400 mg QD Group (N=22) | PF-06826647 50 mg QD->PF-06826647 200 mg QD Group (N=11) | PF-06826647 50 mg QD->PF-06826647 400 mg QD Group (N=11) | PF-06826647 100 mg QD->PF-06826647 200 mg QD Group (N=12) | PF-06826647 100 mg QD->PF-06826647 400 mg QD Group (N=11) | PF-06826647 200 mg QD->PF-06826647 200 mg QD Group (N=45) | PF-06826647 400 mg QD->PF-06826647 400 mg QD Group (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Erythema migrans (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1 | 3 | 1 | 3 | 2 | 6 | 12
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 2 | 0 | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Diffuse axonal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 5 | 6
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 2 | 4 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Prothrombin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Circadian rhythm sleep disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03895372/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT03895372/SAP_001.pdf